CLINICAL TRIAL: NCT02928146
Title: Comparison of Lichtenstein Versus TAPP and TEP Techniques for Inguinal Hernia Repair
Brief Title: Lichtenstein Versus TAPP and TEP in Groin Hernioplasty
Acronym: TAPP&TEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Miroslaw Szura (Other)
Collaborators: Jagiellonian University (Other); Holy Jan Grande Boni Fratres Hospital in Krakow (Unknown); Stefan Zeromski Hospital in Kraków (Unknown)
Responsible Party: Sponsor-Investigator, Miroslaw Szura, Associate Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Lichtenstein vs TAPP/TEP
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Inguinal Hernia
Keywords: TAPP; TEP; Lichtenstein; syntethic mesh; hernioplasty
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lichtenstein technique (Active Comparator): Lichtenstein inguinal hernia repair
  Interventions: Procedure: Hernia Repair
- TAPP (Active Comparator): Transabdominal preperitoneal (TAPP) approach for inguinal hernia repair
  Interventions: Procedure: Hernia Repair
- TEP (Active Comparator): Totally extraperitoneal (TEP) approach for inguinal hernia repair
  Interventions: Procedure: Hernia Repair

INTERVENTIONS:
Procedure: Hernia Repair

SUMMARY:
The aim of the study is to evaluate the effectiveness of various methods of inguinal hernia repair and to evaluate techniques of synthetic mesh fixation during laparoscopic and open hernia repair.

DETAILED DESCRIPTION:
In modern literature there is no conclusive evidence for the superiority of endoscopic over open inguinal hernia repair techniques, due to the lack of prospective, multicenter, randomized studies involving a sufficient number of patients. Both Lichtenstein and TAPP/TEP techniques are widely used and accepted methods of treatment. The clinical significance of this study is to show the differences in the incidence of perioperative complications, the evaluation of postoperative pain, full recovery time and improving the quality of life. The diagnosis of inguinal hernia will be based on a physical examination performed by an experienced surgeon based on the medical history of the patient and, if necessary, on ultrasound examination of the abdominal wall. Random assignment of patients to one of three treatment arms will take place the day before the surgery using computer-generated randomization list. The operating surgeon will be determined prior to randomization. Each patient before the study will receive complete information about the study which will be explained in detail regarding all planned procedures, the patient will obtain answers to any questions. After explaining any doubts the patient will sign the informed consent to participate in the study, in the presence of the investigator. Patients will be divided into three groups - TAPP, TEP and Lichtenstein method. Patients treated by TAPP and Lichtenstein will be further divided into subgroups - fixation glue or stitching - Lichtenstein method; fixation glue, tackers or implantation without fixation - TAPP method. Patients will receive preoperative antibiotic prophylaxis with a single dose of cephalosporin. Patients undergoing surgery will be hospitalized in the Department of Surgery until the first postop day. In justified cases, hospitalization will be extended.

ELIGIBILITY:
Inclusion Criteria:

* male
* age: 18 - 65
* planned inguinal hernia repair using synthetic implant
* BMI range: 20-35 kg / m2
* written informed consent

Exclusion Criteria:

* prior midline laparotomy
* contraindications for general anaesthesia
* ASA > IV
* cirrhosis (Child B or C) or ascites
* active treatment with use of chemiotherapy
* incarcerated hernia

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications associated with wound | 30 days after surgery
  Wound infection with or without the need to remove the mesh, Wound necrosis, Hematoma or seroma in the wound.

SECONDARY OUTCOMES:
The frequency of conversions (from laparoscopic to open approach) | 1 year

OTHER OUTCOMES:
Evaluation of the severity of pain according to VAS (visual analogue scale) | 1 year after surgery
Quality of life. | Prior to surgery, 1 and 6 months after the operation using SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw Szura, MD, PhD, Study Director — Department of Experimental and Clinical Surgery, Jagiellonian University Medical College; Rafal Solecki, MD, PhD, Principal Investigator — Department of Experimental and Clinical Surgery, Jagiellonian University Medical College; Artur Pasternak, MD,PhD, Principal Investigator — Department of Anatomy, Jagiellonian University Medical College; Jakub Łomnicki, MD, Principal Investigator — Stefan Zeromski Hospital in Krakow

IPD SHARING:
Plan to Share IPD: Undecided